CLINICAL TRIAL: NCT06470191
Title: A Multicenter, Randomized, Controlled, Open Phase II/III Clinical Study to Evaluate the Efficacy and Safety of B007 Versus Cyclosporine in the Treatment of Primary Membranous Nephropathy.
Brief Title: A Clinical Study of B007 in the Treatment of Primary Membranous Nephropathy.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPH-B007-302
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-06

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B007 (Experimental)
  Interventions: Drug: B007
- Cyclosporin Capsules (Active Comparator)
  Interventions: Drug: Cyclosporin Capsules

INTERVENTIONS:
Drug: B007 — B007： Subcutaneous injection was administered on days 1 and 15
  Arms: B007
Drug: Cyclosporin Capsules — Cyclosporin Capsules： Orally, 3.5 mg/kg/d；
  Arms: Cyclosporin Capsules

SUMMARY:
To evaluate the efficacy and safety of B007 in the Treatment of Primary Membranous Nephropathy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with primary membranous nephropathy pathologically confirmed by renal biopsy;
2. Subjects with glomerular filtration rate（eGFR） ≥ 45 mL/min/1.73 m2.
3. If taking Angiotensin converting enzyme inhibitors/angiotensin II receptor antagonists/sodium-glucose cotransporter 2 inhibitors/endothelin inhibitors, a stable dose within 4 weeks before randomization;
4. Subjects with 24-hour elevated urinary protein in accordance with the prescribed conditions;
5. Subjects whose laboratory test results meet the prescribed standards during the screening period;
6. Subjects who have fully understood this study and voluntarily signed the informed consent form；
7. Subjects who are able to follow the study protocol as judged by the investigator.

Exclusion Criteria:

1. Subjects with secondary membranous nephropathy or primary membranous nephropathy whose pathological reports suggest concomitant crescent bodies;
2. Subjects identified by the investigator as previously resistant to CD20 monoclonal antibody or cyclosporine;
3. Subjects who have received medication prescribed for membranous nephropathy;
4. Subjects with concomitant prescribed diseases;
5. Subjects with a known history of severe allergic reactions to humanized monoclonal antibodies, or known allergies to any component of cyclosporine or B007;
6. Subjects who received live vaccination, major surgery, or participated in other clinical trials within 28 days before receiving the study drug;
7. Subjects with positive hepatitis B surface antigen; those with positive hepatitis C virus antibody; those with a history of immunodeficiency or suffer from other acquired or congenital immunodeficiency diseases;
8. Subjects who have a clear history of tuberculosis or have received anti-tuberculosis treatment;
9. Subjects with CD4+ T lymphocyte count < 400 cells/μL;
10. Pregnant or lactating women; women of childbearing potential who have not been sterilized do not agree to use appropriate contraceptive measures during treatment and for at least 12 months after the last dose of the study drug;
11. For male subjects who have not been sterilized: those who do not consent to the use of barrier contraception during the study period and for at least 12 months after the last administration of the study drug, and who do not consent to the use of other contraceptive methods by their spouses;
12. Other conditions unsuitable for participation in this study determined by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR（Overall Remission Rate） | Approximately 2 years

SECONDARY OUTCOMES:
CRR（Complete Remission Rate） | Approximately 2 years
PRR（Partial Remission Rate） | Approximately 2 years
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking university first hospital, Beijing
  - The Second Norman Bethune Hospital of Jilin University, Changchun
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - Sir Run Run Shaw Hospital , affiliated with the Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Shandong Provincial Hospital, Jinan
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Affiliated Hospital of Nantong University, Nantong
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Northern Theater Command General Hospital, Shenyang
  - Shengjing Hospital affiliated to China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Xi'an Daxing Hospital, Xi'an
  - The Second Affiliated Hospital of Xingtai Medical college, Xingtai
  - Northern Jiangsu People's Hospital, Yangzhou
  - Yantai Yuhuangding Hospital, Yantai
  - The First People's Hospital of Zigong, Zigong